CLINICAL TRIAL: NCT04161053
Title: Clinical Study Evaluating the Efficacy and Safety of Nitazoxanide in Preventing Recurrence of Hepatic Encephalopathy
Brief Title: Efficacy and Safety of Nitazoxanide in Preventing Recurrence of Hepatic Encephalopathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Encephalopathy
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin; nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin (Active Comparator): 550 mg Rifaximin tablets twice daily for six months.
  Interventions: Drug: Rifaximin
- Nitazoxanide (Experimental): 500 mg Nitazoxanide tablets twice daily for six months.
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 550 mg twice daily for 6 months
  Other Names: Gastrobiotic, Trencedia
  Arms: Rifaximin
Drug: Nitazoxanide — Nitazoxanide 500 mg twice daily for 6 months
  Other Names: Nanazoxid
  Arms: Nitazoxanide

SUMMARY:
Efficacy and Safety of Nitazoxanide in preventing recurrence of Hepatic Encephalopathy.

DETAILED DESCRIPTION:
Clinical Study Evaluating the Efficacy and Safety of Nitazoxanide in preventing recurrence of Hepatic Encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patient with at least one previous episode of hepatic encephalopathy.
* Adult Patients aging from 20 to 65 years old

Exclusion Criteria:

* Active GIT bleeding.
* Major psychiatric illness (psychosis & epilepsy).
* Renal insufficiency (S.Cr 2mg/dl).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of encephalopathy episodes during treatment | 6 months
  The number of encephalopathy episodes during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Khadija Ahmed Glal, Msc, Principal Investigator — Tanta University; Tarek Mohamed Mostafa, ass, Prof., Principal Investigator — Tanta University; Sherief Abd-Elsalam, Ass. Prof., Principal Investigator — Tanta University - Tropical Medicine Department
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No